CLINICAL TRIAL: NCT01903213
Title: Post-Marketing Surveillance on Long-Term Drug Use of Kiklin (Bixalomer)® Capsules in Patients With Hyperphosphatemia Receiving Peritoneal Dialysis
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: KIK002
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2020-03

CONDITIONS: Chronic Renal Failure
Keywords: Peritoneal dialysis; Bixalomer; Chronic renal failure patients with Hyperphosphatemia; Kiklin®
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — bixalomer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kiklin group: Oral
  Interventions: Drug: bixalomer

INTERVENTIONS:
Drug: bixalomer — Oral
  Other Names: Kiklin; ASP1585; AMG223; ILY101

SUMMARY:
To evaluate the safety and efficacy of long-term use of Kiklin® Capsules in actual clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure patients with Hyperphosphatemia receiving peritoneal dialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Chronic renal failure with Hyperphosphatemia receiving Peritoneal dialysis
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2013-03-19 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the incidence of adverse events (including adverse drug reactions), vital signs and laboratory tests | Baseline and 1, 2, 3, 6, 12 months after administration

SECONDARY OUTCOMES:
Serum phosphorous levels | Baseline and 1, 2, 3, 6, 12 months after administration
Serum albumin level | Baseline and 1, 2, 3, 6, 12 months after administration
Serum calcium level | Baseline and 1, 2, 3, 6, 12 months after administration
Serum intact PTH (parathyroid hormone) level | Baseline and 1, 2, 3, 6, 12 months after administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.